CLINICAL TRIAL: NCT04144569
Title: the Effectiveness and Safety Study on PD-1 Combined With Pyrotinib for First-line Chemotherapy Failed HER2 Insertion Mutation Advanced Non-small Cell Lung Cancer
Brief Title: PD-1 Combined With Pyrotinib for Chemotherapy Failure HER2 Insertion Mutation Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POETHIS
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HER2 Insertion Mutation Positive Advanced NSCLC
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Combined With Pyrotinib (Experimental): PD-1 combined With pyrotinib used fo first-line chemotherapy failedr HER2 Insertion mutation positive advanced NSCLC
  Interventions: Drug: PD-1 Combined With Pyrotinib

INTERVENTIONS:
Drug: PD-1 Combined With Pyrotinib — PD-1 Combined With Pyrotinib

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of PD-1 Combined With Pyrotinib for First-line chemotherapy failed HER2 Insertion Mutation Positive Advanced Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced non-small cell lung cancer confirmed by histology or cytology
* HER2 insertion mutation-positive
* Failure with first-line standard chemotherapy
* with measurable lesions.

Exclusion Criteria:

* no measurable tumor lesions
* Patients received PD-1 or Pyrotinib before

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Approximately 1 years
  Progression free survival

SECONDARY OUTCOMES:
ORR | Approximately 1 years
  To measure the patients's overall response rate
OS | Approximately 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China